CLINICAL TRIAL: NCT06247202
Title: Effect of Smart Phone Delivered Health Education Intervention on Overweight and Obese Schoolchildren's Dietary Habits and Body Composition in the UAE
Brief Title: Effect of Smart Phone Health Education on Overweight and Obese Schoolchildren's Dietary Habits and Body Composition
Acronym: mHealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: University of Sharjah (Other)
Responsible Party: Principal Investigator, Heba Mustafaalsaafin, Principal Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USM/JEPeM/KK/23020205; REC-22-09-05-01 (Other: University of Sharjah)
Record Dates: First submitted 2024-01-07; First posted 2024-02-07 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity | interventions — Telemedicine; Congresses as Topic

STUDY DESIGN:
Intervention Model Description: Participants will be randomly divided into intervention group and control group.
  intervention group will receive smart phone delivered nutrition education while control group will receive paper delivered nutrition education.
Who Masked: Outcomes Assessor
Masking Description: Lab technician who will handle the saliva analysis and the person who will be doing the statistical analysis will be blinded of any data related to the grouping of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in the intervention group will receive smart phone delivered health education in the form of text messages through WhatsApp.
  Interventions: Other: Smart Phone Education (mhealth)
- Control group (Active Comparator): Participants in the control group will receive paper delivered health education in the form of a one time handout.
  Interventions: Other: Paper Education (conventional)

INTERVENTIONS:
Other: Smart Phone Education (mhealth) — Nutrition and Health Education module delivered through m-health approach (smart phones)
  Arms: Intervention group
Other: Paper Education (conventional) — Nutrition and Health Education module delivered through conventional approach (paper)
  Arms: Control group

SUMMARY:
The aim of this study is to investigate the effect of mobile health nutrition education intervention in the changing of dietary habits and body composition of overweight and obese 8-12 years old children in Sharjah, United Arab Emirates and to compare its effectiveness to paper educational intervention among the same age group.

The main questions it aims to answer are:

1. Are there any significant changes in dietary habits, physical activity and body composition among overweight and obese school-age children after three months of mobile health intervention?
2. Is there any significant difference between the effect of smart phone delivered and paper delivered interventions (changes in dietary habits, physical activity and body composition) among overweight and obese school-age children after three months of interventions?
3. Are there any significant changes in the obesity inflammatory panel among overweight and obese school-age children after three months of mobile health intervention?
4. Is there any significant difference in the sustainability of the outcomes between mobile health and paper delivered interventions among overweight and obese school-age children two months after the end of the intervention?
5. Are there any significant changes in nutrition related knowledge among parents of overweight and obese school-age children after three months of intervention?

Participants (children with their parents) will be randomly divided into intervention group and control group. Parents of children from the intervention group will receive two text messages/graphics per week about healthy eating and physical activity (PA) on their mobile phones during the intervention period (3 months). While parents in the control group will receive a one-time printed handout containing the same messages at the beginning of the intervention period.

Assessment of children's anthropometry, dietary intake and physical activity will be evaluated pre and post intervention and one more time after a two months period of maintenance after the end of the intervention. Parents' nutrition knowledge will be evaluated pre and post intervention only. Also, children salivary obesity markers will be measured at baseline and at the end of the intervention period to explore the effects of the intervention on inflammatory markers associated with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Overweight/obese children (over 2 SD based on the WHO Growth Reference (2007)).
* Between 8 - 12 years old.
* Attending school in Sharjah, UAE.

Exclusion Criteria:

* Children on a specific diet.
* Children who have any chronic diseases.

Parents qualify if their children meet the inclusion criteria, they can read and speak in Arabic, they plan to stay in Sharjah for six months from the beginning of the intervention, and they own and use a smart phone.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 146 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Weight | 3 times: before intervention (at 0 months), after intervention (at 3 months), after maintenance (at 5 months)
  Will be measured using a Body Composition Analyzer, and will be measured in Kilograms
Height | 3 times: before intervention (at 0 months), after intervention (at 3 months), after maintenance (at 5 months)
  Will be measured using a standing Stadiometer, and will be measured in Centimetres
Body Mass Index | 3 times: before intervention (at 0 months), after intervention (at 3 months), after maintenance (at 5 months)
  Will be calculated using the weight and height, and will be measured in kg/m^2
Body Fat Mass | 3 times: before intervention (at 0 months), after intervention (at 3 months), after maintenance (at 5 months)
  Will be measured using a Body Composition Analyzer, and will be measured in Kilograms
Fat Free Mass | 3 times: before intervention (at 0 months), after intervention (at 3 months), after maintenance (at 5 months)
  Will be measured using a Body Composition Analyzer, and will be measured in Kilograms
Total Body Water | 3 times: before intervention (at 0 months), after intervention (at 3 months), after maintenance (at 5 months)
  Will be measured using a Body Composition Analyzer, and will be measured in Kilograms
Parents' Knowledge | twice: before intervention (at 0 months) and after intervention (at 3 months).
  Using a valid Nutrition Knowledge Attitude Practice Questionnaire - no scale
Children's Dietary Intake | 3 times: before intervention (at 0 months), after intervention (at 3 months), after maintenance (at 5 months)
  Using 24 Hours' Diet recall (3 days).
Children's Physical Activity | 3 times: before intervention (at 0 months), after intervention (at 3 months), after maintenance (at 5 months)
  Using a valid Physical Activity Questionnaire - no scale
Salivary C-Reactive Protein Concentration | twice: before intervention (at 0 months) and after intervention (at 3 months).
  Concentration in saliva samples will be assessed using Luminex Performance Human Obesity Panel (10-Plex)
Salivary Adiponectin (Acrp30) Concentration | twice: before intervention (at 0 months) and after intervention (at 3 months).
  Concentration in saliva samples will be assessed using Luminex Performance Human Obesity Panel (10-Plex)
Salivary Monocyte Chemoattractant Protein-1 (MCP-1/CCL2) Concentration | twice: before intervention (at 0 months) and after intervention (at 3 months).
  Concentration in saliva samples will be assessed using Luminex Performance Human Obesity Panel (10-Plex)
Salivary Complement Factor D (Adipsin) Concentration | twice: before intervention (at 0 months) and after intervention (at 3 months).
  Concentration in saliva samples will be assessed using Luminex Performance Human Obesity Panel (10-Plex)
Salivary Interleukin 6 (IL-6) Concentration | twice: before intervention (at 0 months) and after intervention (at 3 months).
  Concentration in saliva samples will be assessed using Luminex Performance Human Obesity Panel (10-Plex)
Salivary Interleukin 10 (IL-10) Concentration | twice: before intervention (at 0 months) and after intervention (at 3 months).
  Concentration in saliva samples will be assessed using Luminex Performance Human Obesity Panel (10-Plex)
Salivary Leptin (OB) Concentration | twice: before intervention (at 0 months) and after intervention (at 3 months).
  Concentration in saliva samples will be assessed using Luminex Performance Human Obesity Panel (10-Plex)
Salivary Resistin Concentration | twice: before intervention (at 0 months) and after intervention (at 3 months).
  Concentration in saliva samples will be assessed using Luminex Performance Human Obesity Panel (10-Plex)
Salivary Plasminogen Activator Inhibitor-1 (Serpin E1 / PAI-1) Concentration | twice: before intervention (at 0 months) and after intervention (at 3 months).
  Concentration in saliva samples will be assessed using Luminex Performance Human Obesity Panel (10-Plex)
Salivary Tumour Necrosis Factor alpha (TNF alpha) Concentration | twice: before intervention (at 0 months) and after intervention (at 3 months).
  Concentration in saliva samples will be assessed using Luminex Performance Human Obesity Panel (10-Plex)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sharjah, Sharjah city, United Arab Emirates